CLINICAL TRIAL: NCT00063245
Title: Noninvasive Stimulation of Human Deep Brain Regions With a Magnetic Stimulator
Brief Title: Stimulating Deep Brain Regions With a Magnetic Stimulator
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030231; 03-N-0231
Record Dates: First submitted 2003-06-23; First posted 2003-06-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-04

CONDITIONS: Healthy
Keywords: Motor Cortex; Mood; Reward; Transcranial Magnetic Stimulation; Magnetic Coil; Healthy Volunteer; HV

SUMMARY:
The purpose of this study is to determine whether a special coil designed for magnetic stimulation of areas deep in the brain can affect mood and emotion in healthy volunteers. Researchers hope to better understand how the brain controls mood and motivation and what goes wrong with this process in disease.

For transcranial magnetic stimulation (TMS), a wire coil is held over the scalp. A brief electrical current passes through the coil and creates a magnetic pulse that stimulates the brain.

Eighteen participants, 9 men and 9 women, will be enrolled in this study. They will be assigned to one or both of the following two experiments.

Experiment 1

In this experiment, researchers will test the effectiveness of a new type of wire coil. They will deliver magnetic impulses of varying strength. Approximately 150 stimulations will be given over of about 20 minutes. To determine whether the coil causes any problem with hearing, participants will undergo a hearing test immediately before and after the experiment.

Experiment 2

This experiment, which has two parts, is designed to determine whether TMS can affect mood. In the first part, participants will be asked to report any changes in mood before, during and after the magnetic stimulation. In the second part, they will be asked to choose between sets of 2 identical pictures-choosing one will result in full magnetic stimulation, choosing the other will result in stimulation at 10 percent of full intensity.

Participants will be compensated up to $100 for their involvement in this study.

DETAILED DESCRIPTION:
Current magnetic stimulation techniques permit only superficial stimulation of brain, but for some purposes deeper stimulation would be helpful. The purpose of this study is to determine whether a special coil designed for magnetic stimulation of deep brain regions can affect mood and emotion in healthy human volunteers. The special coil was designed to stimulate neuronal pathways related to the control of motivation and reward, specifically, fibers connecting the cingulated or prefrontal cortex with the nucleus accumbens. Computerized theoretical calculations were made in order to optimize the coil design for maximizing the percentage of stimulation in depth relative to the cortical regions. The present study will look first at the influence of the coil on the response from motor cortex. Should there be good evidence the coil can truly be more effective in stimulating deep structures, then we will explore whether it can indeed affect mood and emotion when single pulses are applied.

ELIGIBILITY:
INCLUSION CRITERIA:

The study is planned for adult subjects with normal neurologic and psychiatric examinations.

Healthy male and female volunteers will be included in this protocol.

EXCLUSION CRITERIA:

History of surgery with metallic implants or known history of metallic particles in the eye, cardiac pacemaker, neurostimulators, cochlear implants, history of drug abuse, psychiatric illness, hypertension, or concurrent medication.

Children are also excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18
Dates: Start 2003-06; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Breiter HC, Rosen BR. Functional magnetic resonance imaging of brain reward circuitry in the human. Ann N Y Acad Sci. 1999 Jun 29;877:523-47. doi: 10.1111/j.1749-6632.1999.tb09287.x. PMID 10415669
- [Background] Breiter HC, Gollub RL, Weisskoff RM, Kennedy DN, Makris N, Berke JD, Goodman JM, Kantor HL, Gastfriend DR, Riorden JP, Mathew RT, Rosen BR, Hyman SE. Acute effects of cocaine on human brain activity and emotion. Neuron. 1997 Sep;19(3):591-611. doi: 10.1016/s0896-6273(00)80374-8. PMID 9331351
- [Background] Eaton H. Electric field induced in a spherical volume conductor from arbitrary coils: application to magnetic stimulation and MEG. Med Biol Eng Comput. 1992 Jul;30(4):433-40. doi: 10.1007/BF02446182. PMID 1487945